CLINICAL TRIAL: NCT05979935
Title: A Clinical Study on the Diagnostic Value of Digital Tongue Diagnosis Model for High- and Low-risk Esophagogastroduodenal Varices in Patients With Liver Cirrhosis
Brief Title: A Digital Tongue Diagnosis Model for High- and Low-risk Esophagogastroduodenal Varices in Cirrhosis
Status: Active, not recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Shanghai Changzheng Hospital (Other); Shanghai East Hospital of Tongji University (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other); Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other); Tianjin Medical University General Hospital (Other); Army Medical Center of PLA (Other Government); Shandong Provincial Hospital (Other Government); Qianfoshan Hospital (Other); Shandong Public Health Clinical Center (Other Government); The 960th Hospital of the PLA Joint Logistics Support Force (Unknown); Jinan Central Hospital (Other); Weifang People's Hospital (Other); Liaocheng People's Hospital (Other); The Second Affiliated Hospital of Shandong First Medical University (Other); Jining First People's Hospital (Other)
Responsible Party: Principal Investigator, Yanjing Gao, Professor, Qilu Hospital of Shandong University
Other Study IDs: 20230726-QiluH
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Esophageal Varices; Liver Cirrhosis; Sublingual Varices; Portal Hypertension
Keywords: Esophagogastroduodenal Varices; Liver cirrhosis; Sublingual vein; Portal hypertension
MeSH Terms: conditions — Esophageal and Gastric Varices; Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with high-risk of esophageal varices in liver cirrhosis: The maximum diameter of varices ≥ 5 mm or maximum diameter of varices <5mm with positive red sign in patients with liver cirrhosis
  Interventions: Diagnostic Test: tongue diagnosis
- patients with low-risk of esophageal varices in liver cirrhosis: the maximum diameter of esophageal varices < 5 mm without positive red sign in patients with liver cirrhosis.
  Interventions: Diagnostic Test: tongue diagnosis

INTERVENTIONS:
Diagnostic Test: tongue diagnosis — The tongue image of participants will be collected via camera, and tongue images will be used for AI deep model learning analysis.

SUMMARY:
The aim of this observational study is to establish an AI deep learning model that can dianosie high-risk varices for patients with cirrhosis effeciently.

The main question of this study is to esplore:

question 1: Developing a digital tongue diagnosis model, specifically a deep learning model to diagnose high-risk esophageal and gastric varices (HRV) associated with cirrhosis using sublingual vein images. Answering the question of whether the new tongue diagnosis method can accurately diagnose.

Question 2: Compare the diagnostic efficacy digital tongue diagnosis model with diagnostic models constructed using other biochemical indicators for HRV in cirrhosis, and answer the question of "how to use it optimally."

Question 3: Exploring the correlation between sublingual vein characteristics and Hepatic venous pressure gradient (HVPG).

Question 4: Compared with endoscopic examination results, validate the diagnostic performance of the model (AUC ≥ 0.90) and screen for key parameters of sublingual vein characteristics (such as sublingual vein varicosity diameter, vein length, color, etc.).

Question 5: Follow-up tongue examination images of patients with cirrhosis who underwent treatment (e.g., endoscopy, splenic embolization, TIPS, etc.) at 1, 2, and 3 years post-treatment were evaluated to assess the efficacy of digital tongue examination models in predicting high-risk esophageal and gastric variceal bleeding at 1, 2, and 3 years post-treatment, as well as the efficacy in predicting endoscopic treatment failure rates and patient mortality associated with bleeding.

DETAILED DESCRIPTION:
Firstly, participants will be divided into two groups according to their degree of esophageal varices from endoscopic examination and CT report, including high-risk varices (HRV) group and low-risk varices (LRV) group. Secondly, participants will be asked to show their tongue, including the surface and sublingual veins of tongue, and the tongue images of each participants will be collected by researchers via camera. After finishing tongue image collection, participants will receive a professional tongue diagnosis report in Traditional Chinese Medicine and health suggestion. Finally, tongue images will be analyzed by AI deep learning model and some specifialized information will be estracted exactly. Besides, 60 patietns will be selected to eplore whtether sublingual vein characteristics is assoicated with HVPG. Finally, patietns will be followed up during 3 years, and gastric variceal bleeding, endoscopic treatment failure rates, and patient mortality risks related to bleeding will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years (including both age limits), no gender restrictions;
2. Diagnosed with cirrhosis based on clinical presentation, laboratory tests, imaging studies, and/or histopathological examination;
3. Undergone upper gastrointestinal endoscopy within the past 3 months prior to enrollment and have complete endoscopic imaging records;
4. Undergone enhanced CT or MRI scan of the upper abdomen within the past month prior to enrollment;
5. Patients who consent to enrollment and have signed an informed consent form.

Exclusion Criteria:

1. Patients who have previously undergone endoscopic treatment for esophageal or gastric varices, transjugular intrahepatic portosystemic shunt (TIPS), splenectomy, hepatectomy, balloon occlusion of the portal vein, or liver transplantation;
2. Patients with grade 2-3 ascites or overt hepatic encephalopathy;
3. Patients with a history of portal venous system thrombosis (including the portal vein, splenic vein, superior mesenteric vein, etc.) or portal venous cavernous transformation, and who have been diagnosed with thrombosis within the past two weeks;
4. Patients diagnosed with or suspected of having primary liver cancer or other advanced malignant tumors;
5. Patients with chronic obstructive pulmonary disease and right heart failure;
6. Male and female patients with moderate anemia (hemoglobin <70 g/L);
7. Patients with poorly controlled diabetes or microvascular complications;
8. Patients with poorly controlled hypertension;
9. Patients with hematological disorders such as polycythemia vera;
10. Patients with local oral lesions affecting sublingual venous blood flow, such as Ludwig's angina, Lemierre syndrome, or complications following certain oral surgeries (e.g., scar contracture or hematoma after tongue or floor of mouth surgery);
11. Patients with sublingual venous varicosities;
12. Patients who have experienced other severe systemic infections within the past 2 weeks prior to enrollment;
13. Pregnant women and peripartum women;
14. Patients with mental disorders;
15. Patients with incomplete medical records;
16. Patients unable to cooperate in completing the clinical study;
17. Other reasons deemed unsuitable for participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects in this study are patients with liver cirrhosis from the Department of Gastroenterology, Qilu Hospital, Shandong University and other 15 hospitaals. According to the 《Prevention and Treatment Plan for Viral Hepatitis》 revised by the Infectious Diseases and Parasitic disease Branch and Hepatology Branch of the Chinese Medical Association in September 2000, Patients with liver cirrhosis and esophageal varices aged 18-75 years will be included in the study.
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
AUC of tongue diagnostic model | through study completion, up to 3 years
  Using endoscopic diagnostic criteria as the "gold standard," we calculated the area under the ROC curve (AUC), sensitivity, specificity, positive predictive value, and negative predictive value of the VIT-based digital tongue diagnosis model to evaluate its diagnostic performance in diagnosing HRV in cirrhosis.

SECONDARY OUTCOMES:
ROC of biochemical characteristic | through study completion, up to 3 years
  Calculate the AUC valthe digital tongue diagnosis model.ue, sensitivity, specificity, positive predictive value, negative predictive value, and other relevant parameters of the ROC curve for the HRV diagnostic model for cirrhosis constructed based on biochemical indicators, and compare them with
Association between HVPG and sublingual vein | through study completion, up to 3 years
  The association between sublingual vein and HVPG
Characteristic of sublingual vein | through studyy completion, up to 3 years
  Key parameters for screening sublingual vein characteristics (such as sublingual vein varicosity diameter, vein length, color, etc.).
The rate of esophageal variceal bleeding, endoscopic treatment failure, and patient mortality | through study completion, up to 3 years
  The incidence of esophageal variceal bleeding, endoscopic treatment failure rate, and patient mortality related to bleeding in patients with cirrhosis 1, 2, and 3 years after diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Yanjing Gao, PhD MD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shdong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ou J, Li R, Zeng R, Wu CQ, Chen Y, Chen TW, Zhang XM, Wu L, Jiang Y, Yang JQ, Cao JM, Tang S, Tang MJ, Hu J. CT radiomic features for predicting resectability of oesophageal squamous cell carcinoma as given by feature analysis: a case control study. Cancer Imaging. 2019 Oct 16;19(1):66. doi: 10.1186/s40644-019-0254-0. PMID 31619297
- [Result] Tandon M, Singh H, Singla N, Jain P, Pandey CK. Tongue thickness in health vs cirrhosis of the liver: Prospective observational study. World J Gastrointest Pharmacol Ther. 2020 Aug 8;11(3):59-68. doi: 10.4292/wjgpt.v11.i3.59. PMID 32844044
- [Result] He C, Liao Q, Fu P, Li J, Zhao X, Zhang Q, Gui Q. Microbiological characteristics of different tongue coatings in adults. BMC Microbiol. 2022 Sep 9;22(1):214. doi: 10.1186/s12866-022-02626-7. PMID 36085010
- [Result] Lin Y, Li L, Yu D, Liu Z, Zhang S, Wang Q, Li Y, Cheng B, Qiao J, Gao Y. A novel radiomics-platelet nomogram for the prediction of gastroesophageal varices needing treatment in cirrhotic patients. Hepatol Int. 2021 Aug;15(4):995-1005. doi: 10.1007/s12072-021-10208-4. Epub 2021 Jun 11. PMID 34115257
- [Result] Gralnek IM, Camus Duboc M, Garcia-Pagan JC, Fuccio L, Karstensen JG, Hucl T, Jovanovic I, Awadie H, Hernandez-Gea V, Tantau M, Ebigbo A, Ibrahim M, Vlachogiannakos J, Burgmans MC, Rosasco R, Triantafyllou K. Endoscopic diagnosis and management of esophagogastric variceal hemorrhage: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2022 Nov;54(11):1094-1120. doi: 10.1055/a-1939-4887. Epub 2022 Sep 29. PMID 36174643
- [Result] de Franchis R, Bosch J, Garcia-Tsao G, Reiberger T, Ripoll C; Baveno VII Faculty. Baveno VII - Renewing consensus in portal hypertension. J Hepatol. 2022 Apr;76(4):959-974. doi: 10.1016/j.jhep.2021.12.022. Epub 2021 Dec 30. PMID 35120736